CLINICAL TRIAL: NCT01435577
Title: A Randomized, Double-blind, Placebo-controlled Parallel Group, Multicenter Trial to Evaluate the Efficacy and Safety of Multiple Dose Administration of an Intravenous Formulation of Tapentadol in the Treatment of Acute Pain Following Bunionectomy.
Brief Title: Intravenous Tapentadol in Post-Bunionectomy Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 295054
Record Dates: First submitted 2011-09-15; First posted 2011-09-16 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Bunion; Pain
Keywords: Bunionectomy; Postsurgical Pain; Acute Pain
MeSH Terms: conditions — Bunion; Pain; Pain, Postoperative; Acute Pain | interventions — Tapentadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tapentadol intravenous (Experimental): Tapentadol will be given by intravenous infusion. Tapentadol will be administered every 4 hours. Ibuprofen 600 mg orally may be given as rescue medication for pain not controlled by Tapentadol alone.
  Interventions: Drug: Tapentadol
- Matching placebo intravenous (Placebo Comparator): Placebo (0.9% sodium chloride and water for injection). Ibuprofen 600 mg orally may be given as rescue medication for pain.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Tapentadol — 30 mg per administration, maximum 12 administrations over 48 hours
  Other Names: Palexia, Nucynta
  Arms: Tapentadol intravenous
Drug: Matching Placebo — Maximum 12 administrations over 48 hours
  Arms: Matching placebo intravenous

SUMMARY:
The purpose of this trial is to established the safety and efficacy of multiple dose treatment with tapentadol IV in an adult population with moderate to severe pain following bunionectomy.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo primary unilateral first metatarsal bunionectomy
* Female patients must be postmenopausal, surgically sterile, or practicing an effective method of birth control if they are sexually active
* Qualifying pain intensity (within a maximum of 5 hours after the last surgical stitch) and Baseline pain intensity (last pain score measured within 10 minutes before dosing) 5 on an 11-point (0 to 10) pain intensity numerical rating scale (NRS).

Exclusion Criteria:

* History of malignancy within the past 2 years
* Current or history of alcohol or drug abuse.
* Clinically relevant pulmonary, gastrointestinal, endocrine, metabolic, neurological, psychiatric disorders (resulting in disorientation, memory impairment or inability to report accurately
* History of seizure disorder, epilepsy, or any condition that would put the subject at risk of seizures
* Severely impaired renal function
* Moderately or severely impaired hepatic function
* Contraindications, or a history of allergy or hypersensitivity, to tapentadol, ibuprofen, or excipients
* Use of prohibited concomitant medication, or not allowed use of restricted concomitant medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this trial was from the 26 September 2011 and was completed on the 14 Feb 2012.
Pre-assignment Details: 177 participants signed informed consent.
  * 132 participants underwent surgery.
  * 131 participants reported a pain intensity that qualified them to enter the trial, i.e. one participant did not report sufficient pain to enter the trial.
  * 129 participants were randomized to receive treatment.
Groups:
- Tapentadol Intravenous: Tapentadol will be given by intravenous infusion. Tapentadol will be administered every 4 hours. Ibuprofen 600 mg orally may be given as rescue medication for pain not controlled by tapentadol alone.
  64 Participants Randomized, 64 Participants in the Safety Set (SAF), 64 Participants in the Full Analysis Set (FAS). The FAS comprised all randomized subjects who were administered at least 1 dose and had a baseline pain assessment.
- Matching Placebo Intravenous: Placebo (0.9% sodium chloride and water for injection). Ibuprofen 600 mg orally may be given as rescue medication for pain.
  65 Randomized participants, 65 Participants in the Safety Set (SAF), 65 Participants in the Full Analysis Set(FAS). The FAS comprised all randomized subjects who were administered at least 1 dose and had a baseline pain assessment.
Period: Overall Study
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous
Started | 64 | 65
Completed | 47 | 13
Not Completed | 17 | 52
Not completed — Adverse Event | 10 | 0
Not completed — Lack of Efficacy | 7 | 51
Not completed — Alternative treatment started | 0 | 1

BASELINE CHARACTERISTICS:
Population: The summary statistics provided for baseline was based on safety population that included 64 subjects in the tapentadol group and 65 in the placebo group. The safety population includes randomized participants that received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous | Total
Number analyzed (Participants) | 64 | 65 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (12.61) | 35.8 (12.41) | 38.5 (12.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 60 | 117
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 64 | 65 | 129
Baseline pain intensity [Mean (Standard Deviation); unit: units on a scale] — Pain intensity assessed prior to the first administration of study medication. Pain intensity is assessed by the participant using an 11-point Numeric rating scale (NRS) where a score of zero indicates "no pain" and a score of ten indicates "pain as bad as you can imagine".
  units on a scale | 7.2 (1.41) | 7.3 (1.54) | 7.2 (1.47)

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Differences (SPID 24)
Description: Pain Intensity assessed at predefined time points (at 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 20 and 24 hours after first drug administration) over a 24 hour period using an 11-point Numeric Rating Scale (NRS) where a score of zero indicates "no pain" and a score of ten indicates "pain as bad as you can imagine". Pain Intensity Differences at each predefined time point (calculated as post-baseline NRS values - baseline NRS values) were analyzed. Negative SPID24 values indicate a decrease in pain intensity and positive values indicate an increase in pain intensity since baseline.
Time Frame: Baseline value; up to 24 hours after first study drug administration
Population: Full Analysis Set (FAS): patients who took at least one dose of study medication, had a baseline value, and had at least one post-baseline measurement; Last Observation Carried Forward (LOCF) after dropout, and LOCF for 6 hours after each rescue medication intake.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous
Number analyzed (Participants) | 64 | 65
units on a scale | -51.23 [-59.93 to -42.52] | 25.46 [16.82 to 34.10]

2. Secondary Outcome: Mean Pain Intensity Scores at Fixed Time Points
Description: The mean pain intensity at fixed time points in the trial for all participants is listed. The pain intensity was measured using the Pain Intensity (PI). Pain intensity was assessed on 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine.
Time Frame: Baseline; up to 48 hours
Population: Full Analysis Set (FAS). Participants who took at least one dose of study medication, had a baseline value, and had at least one post-baseline measurement; Last Observation Carried Forward (LOCF) after dropout, and LOCF for 6 hours after each rescue medication intake.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous
Number analyzed (Participants) | 64 | 65
units on a scale
  Baseline (before first study drug administration) | 7.2 (1.41) | 7.3 (1.54)
  0.25 hours after first dose | 3.7 (1.99) | 7.1 (1.57)
  0.5 hour after first dose | 3.1 (1.77) | 7.4 (1.63)
  1 hour after first dose | 3.6 (1.77) | 7.8 (1.76)
  2 hours after first dose | 5.8 (2.03) | 8.5 (1.5)
  4 hours after first dose | 6.1 (1.92) | 8.6 (1.46)
  6 hours after first dose | 6.3 (2.25) | 8.7 (1.47)
  8 hours after first dose | 6.5 (2.29) | 8.6 (1.61)
  12 hours after first dose | 5.2 (2.7) | 8.5 (1.67)
  16 hours after first dose | 3.8 (2.58) | 8.2 (2.12)
  20 hours after first dose | 3.7 (2.52) | 8.0 (2.24)
  24 hours after first dose | 4.1 (2.43) | 8.1 (2.08)
  36 hours after first dose | 3.9 (2.49) | 8.0 (2.39)
  48 hours after first dose | 4.3 (2.56) | 8.1 (2.21)

3. Secondary Outcome: Pain Intensity Differences at Fixed Time Points
Description: Pain Intensity (PI) was assessed on 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine. Pain Intensity Difference (PID) was the difference between baseline pain intensity (prior to the first dose) and the pain intensity at the time. A negative number indicates a decrease in pain in the whole treatment group. The greater the negative pain intensity difference value the greater the pain relief in the treatment arm. A score of 0 indicates that there has been no change in pain in a treatment group. A positive value indicates an increase in pain in the treatment group.
Time Frame: Starting at 15 minutes and up to 48 hours after first drug administration
Population: Full Analysis Set (FAS): Participants who took at least one dose of study medication, had a baseline value, and had at least one post-baseline measurement; Last Observation Carried Forward (LOCF) after dropout, and LOCF for 6 hours after each rescue medication intake.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous
Number analyzed (Participants) | 64 | 65
units on a scale
  0.25 hours after first administration | -3.5 (2.22) | -0.2 (0.95)
  0.5 hours after first administration | -4.1 (2.24) | 0.1 (1.18)
  1 hour after first administration | -3.5 (2.07) | 0.5 (1.4)
  2 hours after first administration | -1.3 (2.24) | 1.2 (1.39)
  4 hours after first dose administration | -1.0 (2.09) | 1.4 (1.47)
  6 hours after first dose administration | -0.9 (2.32) | 1.4 (1.51)
  8 hours after first dose administration | -0.7 (2.5) | 1.3 (1.58)
  12 hours after first dose administration | -2.0 (3.01) | 1.2 (1.57)
  16 hours after first dose administration | -3.4 (2.90) | 0.9 (1.82)
  20 hours after first dose administration | -3.5 (2.89) | 0.7 (2.08)
  24 hours after first dose administration | -3.1 (2.65) | 0.9 (2.0)
  36 hours after first dose administration | -3.2 (2.68) | 0.8 (2.26)
  48 hours after first dose administration | -2.9 (2.76) | 0.8 (2.11)

4. Secondary Outcome: Patient Global Impression of Change After 12 Hours of Treatment
Description: In the Patient Global Impression of Change (PGIC) the participant indicates the perceived change over the treatment period. The participant verbally rated their impression of overall status with 1 of 7 possible responses (very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse).
Time Frame: Baseline value to 12 hours after first study drug administration
Population: Participants contributing data. Missing PGIC values were mainly due to participants discontinuing the trial before this time point.
Measure: Number; unit: participants
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous
Number analyzed (Participants) | 54 | 15
participants
  Very Much Improved | 11 | 0
  Much Improved | 20 | 1
  Minimally Improved | 14 | 9
  No Change | 5 | 4
  Minimally Worse | 4 | 1
  Much Worse | 0 | 0
  Very Much Worse | 0 | 0

5. Secondary Outcome: Patients Global Impression of Change After 24 Hours of Treatment
Description: as for outcome 4
Time Frame: Baseline value to 24 hours after study drug administration
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous
Number analyzed (Participants) | 52 | 15
participants
  Very Much Improved | 13 | 0
  Much Improved | 26 | 5
  Minimally Improved | 11 | 6
  No Change | 1 | 2
  Minimally Worse | 1 | 2

6. Secondary Outcome: Patient Global Impression of Change After 48 Hours of Treatment
Description: as for outcome 4
Time Frame: Baseline value to 48 hours after first study drug administration
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous
Number analyzed (Participants) | 47 | 13
participants
  Very Much Improved | 19 | 2
  Much Improved | 24 | 8
  Minimally Improved | 4 | 2
  No Change | 0 | 1
  Minimally Worse | 0 | 0
  Much Worse | 0 | 0
  Very Much Worse | 0 | 0

7. Secondary Outcome: Sum of Pain Intensity Differences After 60 Minutes
Description: Pain Intensity (PI) was assessed on 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine. Pain Intensity Difference (PID) was the difference between the PI after fixed times after first dose and the baseline PI (prior to the first dose). The Sum of Pain Intensity Differences over 60 minutes was calculated. If the value is negative then the baseline pain intensity was greater than the pain intensity measured after dosing.
Time Frame: Baseline value to 60 minutes after first study drug administration
Population: Full analysis set.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous
Number analyzed (Participants) | 64 | 65
units on a scale | -3.65 [-4.01 to -3.3] | 0.26 [-0.10 to 0.61]

8. Secondary Outcome: Sum of Pain Intensity Differences After 4 Hours
Description: Pain Intensity (PI) was assessed on 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine. Pain Intensity Difference (PID) was the difference between the PI after fixed times after first dose and the baseline PI (prior to the first dose). The Sum of Pain Intensity Differences over 4 hours was calculated. If the values are negative (then the baseline pain intensity was greater than the pain intensity measured after dosing).
Time Frame: Baseline value to 4 hours after first study drug intake
Population: Full analysis set. Primary imputation method was analyzed: Last Observation Carried Forward (LOCF) after dropout, and LOCF for 6 h after each rescue medication intake.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous
Number analyzed (Participants) | 64 | 65
units on a scale | -6.76 [-7.92 to -5.61] | 4.22 [3.07 to 5.37]

9. Secondary Outcome: Sum of Pain Intensity Differences After 8 Hours
Description: Pain Intensity (PI) was assessed on 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine. Pain Intensity Difference (PID) was the difference between the PI after fixed times after first dose and the baseline PI (prior to the first dose). The Sum of Pain Intensity Differences over 8 hours was calculated. If the values are negative (then the baseline pain intensity was greater than the pain intensity measured after dosing).
Time Frame: Baseline value to 8 hours after first study drug administration
Population: Full Analysis Set.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous
Number analyzed (Participants) | 64 | 65
units on a scale | -9.9 [-12.5 to -7.31] | 9.74 [7.17 to 12.32]

10. Secondary Outcome: Sum of Pain Intensity Differences After 12 Hours
Description: Pain Intensity (PI) was assessed on 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine. Pain Intensity Difference (PID) was the difference between the PI after fixed times after first dose and the baseline PI (prior to the first dose). The Sum of Pain Intensity Differences over 12 hours was calculated. If the values are negative (then the baseline pain intensity was greater than the pain intensity measured after dosing).
Time Frame: Baseline value to 12 hours after first study drug administration
Population: Full Analysis Set.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous
Number analyzed (Participants) | 64 | 65
units on a scale | -14.98 [-19.09 to -10.87] | 14.82 [10.74 to 18.90]

11. Secondary Outcome: Sum of Pain Intensity Differences After 48 Hours
Description: Pain Intensity (PI) was assessed on 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine. Pain Intensity Difference (PID) was the difference between the PI after fixed times after first dose and the baseline PI (prior to the first dose). The Sum of Pain Intensity Differences over 60 minutes was calculated. If the values are negative (then the baseline pain intensity was greater than the pain intensity measured after dosing).
Time Frame: Baseline value to 48 hours after first study drug administration
Population: Full Analysis Set.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous
Number analyzed (Participants) | 64 | 65
units on a scale | -122.93 [-143.73 to -102.13] | 45.86 [25.22 to 66.5]

12. Secondary Outcome: Number of Participants With 30% Response After 12 Hours, Based on Pain Intensity Scores
Description: Individual participant response. Number of participants that reported a 30% or more reduction in pain intensity from the administration of the first dose to 12 hours after the first study drug administration are counted as having a response if their pain intensity decreased by 30% from their baseline value.
Time Frame: Baseline value to 12 hours after first study drug administration
Population: Full analysis set.
Measure: Number; unit: participants
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous
Number analyzed (Participants) | 64 | 65
participants | 27 | 1

13. Secondary Outcome: Number of Participants With 30% Response After 24 Hours, Based on Pain Intensity Scores
Description: Individual participant response. Number of participants that reported a 30% or more reduction in pain intensity from the administration of the first dose to 24 hours after the first study drug administration are counted as having a response if their pain intensity decreased by 30% from their baseline value.
Time Frame: Baseline value to 24 hours after first study drug administration
Population: Full analysis set.
Measure: Number; unit: participants
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous
Number analyzed (Participants) | 64 | 65
participants | 31 | 4

14. Secondary Outcome: Number of Participants With 30% Response After 48 Hours, Based on Pain Intensity Scores
Description: Individual participants response. Number of participants that reported a 30% or more reduction in pain intensity from the administration of the first dose to 48 hours after the first study drug administration are counted as having a response if their pain intensity decreased by 30% from their baseline value.
Time Frame: Baseline value to 48 hours after first study drug administration
Population: Full analysis set.
Measure: Number; unit: participants
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous
Number analyzed (Participants) | 64 | 65
participants | 8 | 1

15. Secondary Outcome: Number of Participants With 50% Response After 12 Hours, Based on Pain Intensity Scores
Description: Individual participant response. Number of participants that reported a 50% or more reduction in pain intensity from the administration of the first dose to 12 hours after the first study drug administration are counted as having a response if their pain intensity decreased by 50% from their baseline value.
Time Frame: Baseline value to 12 hours after first study drug administration
Population: Full analysis set.
Measure: Number; unit: participants
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous
Number analyzed (Participants) | 64 | 65
participants | 18 | 1

16. Secondary Outcome: Number of Participants With 50% Response After 24 Hours, Based on Pain Intensity Scores
Description: Individual participant response. Number of participants that reported a 50% or more reduction in pain intensity from the administration of the first dose to 24 hours after the first study drug administration are counted as having a response if their pain intensity decreased by 50% from their baseline value.
Time Frame: Baseline value to 24 hours after first study drug administration
Population: Full analysis set.
Measure: Number; unit: participants
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous
Number analyzed (Participants) | 64 | 65
participants | 24 | 1

17. Secondary Outcome: Number of Participants With 50% Response After 48 Hours, Based on Pain Intensity Scores
Description: Individual participant response. Number of participants that reported a 50% or more reduction in pain intensity from the administration of the first dose to 48 hours after the first study drug administration are counted as having a response if their pain intensity decreased by 50% from their baseline value.
Time Frame: Baseline value to 48 hours after first study drug administration
Population: Full analysis set.
Measure: Number; unit: participants
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous
Number analyzed (Participants) | 64 | 65
participants | 6 | 0

18. Secondary Outcome: Time to First Rescue Medication
Description: The median time to first rescue medication intake (600 mg ibuprofen) in hours.
Time Frame: up to 48 hours
Population: Full analysis set.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous
Number analyzed (Participants) | 64 | 65
hours | 5.4 [4.7 to 7.1] | 2.1 [1.9 to 2.3]

19. Secondary Outcome: Time to Perceptible Pain Relief
Description: When the participant began to feel any pain-relieving effect after the administration of the first dose they were requested to stop the first stopwatch. The time was noted. This measured when the participant first felt any difference in the pain.
Time Frame: up to 48 hours
Population: Participants without pain relief (as measured by the double stopwatch method) were censored at 12 hours from the initial dose or at the time of early withdrawal from the Double-blind Treatment Period, whichever occurred first. Time to perceptible pain relief is not reported for matching placebo arms because of the high number of discontinuations.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Tapentadol Intravenous
Number analyzed (Participants) | 65
hours | 0.2 [0.1 to 0.2]

20. Secondary Outcome: Time to Meaningful Pain Relief
Description: The participant was instructed to stop the stopwatch when they had meaningful pain relief. That is, when the pain relief made a real difference, after the first drug administration.
Time Frame: up to 48 hours
Population: Participants without pain relief (as measured by the double stopwatch method) were censored at 12 hours from the initial dose or at the time of early withdrawal from the Double-blind Treatment Period, whichever occurred first. Time in hours to meaningful pain relief are not reported for matching placebo arm due to the high discontinuation rate.
Measure: Median (95% Confidence Interval); unit: hours
Groups:
- Tapentadol Intravenous: Tapentadol will be given by intravenous infusion. Tapentadol will be administered every 4 hours. Ibuprofen 600 mg orally may be given as rescue medication for pain not controlled by tapentadol alone. Values collected after 12 hours were censored, i.e. participants scored as having no meaningful pain relief.
Arm/Group | Tapentadol Intravenous
Number analyzed (Participants) | 64
hours | 0.3 [0.3 to 0.4]

21. Secondary Outcome: Pharmacokinetic Concentrations of Tapentadol
Description: Tapentadol concentrations were measured in participants in the tapentadol treatment arm. Serum was analyzed by means of liquid chromatography coupled to tandem mass spectrometry with a lower limit of quantification (LLOQ) at 0.2 ng/mL.
Time Frame: 15 minutes to 20 hours after first drug administration
Population: Participants in the placebo arm were not analyzed. Only those participants contributing data were analyzed. Participants that had an early second study drug administration were not part of the analysis.
Measure: Mean (Full Range); unit: ng/mL
Groups:
- Tapentadol Intravenous: Pharmacokinetic samples were taken from all participants, however only samples from the tapentadol treatment group were analyzed.
Arm/Group | Tapentadol Intravenous
Number analyzed (Participants) | 17
ng/mL
  15 minutes after first infusion | 201.2 [69.5 to 593]
  30 minutes after first infusion | 99.5 [59.8 to 164]
  60 minutes after first infusion | 76.4 [43.3 to 103]
  4 hours after end of first infusion: number analyzed (Participants) | 13
  4 hours after end of first infusion | 38.2 [21.5 to 60.5]
  3.5 hours after end of fifth infusion: number analyzed (Participants) | 13
  3.5 hours after end of fifth infusion | 73.2 [39.4 to 106]
  4 hours after end of fifth infusion: number analyzed (Participants) | 9
  4 hours after end of fifth infusion | 70.3 [34.4 to 105]

22. Post Hoc Outcome: Number of Participants Scored as a Responder Based on Patient Global Impression of Change
Description: Responders are those participants with Patient Global Impression of Change (PGIC) values "Much improved", or "Very much improved". Participants with missing value are considered non-responders.
Time Frame: Fixed time points at 12, 24 and 48 hours after baseline
Population: Participants with early second dose the PGIC assessment from End-of-double-blind Treatment was taken as the 48 hours value. Assessments done more than 4.5 hours after the 12th infusion were excluded from analysis and participants were considered non-responders.
Measure: Number; unit: participants
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous
Number analyzed (Participants) | 64 | 65
participants
  Responders 12 hours after first dose | 31 | 1
  Responders 24 hours after first dose | 39 | 5
  Responders 48 hours after first dose | 43 | 10

23. Secondary Outcome: Pharmacokinetic Concentrations of Tapentadol-O-glucuronide
Description: Tapentadol-O-glucuronide is the metabolite of tapentadol. Metabolites are sometimes referred to as "breakdown products". The body alters the administered medication to a metabolite so that can be more easily or quickly removed from the body. Tapentadol-O-glucuronide concentrations were measured in participants in the tapentadol treatment arm. Serum was analyzed by means of liquid chromatography coupled to tandem mass spectrometry with a lower limit of quantification (LLOQ) at 0.2 ng/mL.
Time Frame: 15 minutes to 20 hours after first drug administration
Population: as for outcome 21
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Tapentadol Intravenous
Number analyzed (Participants) | 17
ng/mL
  15 minutes after first infusion: number analyzed (Participants) | 15
  15 minutes after first infusion | 26.4 [11.6 to 88.2]
  30 minutes after first infusion | 290.4 [111 to 515]
  60 minutes after first infusion | 488.2 [287 to 666]
  4 hours after end of first infusion: number analyzed (Participants) | 13
  4 hours after end of first infusion | 452.4 [265 to 651]
  3.5 hours after end of fifth infusion: number analyzed (Participants) | 13
  3.5 hours after end of fifth infusion | 1048.7 [680 to 1410]
  4 hours after end of fifth infusion: number analyzed (Participants) | 9
  4 hours after end of fifth infusion | 945.1 [608 to 1200]

24. Secondary Outcome: Mean Pain Intensity Scores at Relative Time- Tapentadol Randomized Participants
Description: The pain intensity at the relative time points are the pain intensity before and one hour after study drug administration. The pain intensity was measured using the Pain Intensity (PI). Pain intensity was assessed on 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine.
Time Frame: Baseline; for the first 6 administrations
Population: Participants contributing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Intravenous
Number analyzed (Participants) | 64
units on a scale
  Prior to first dose (n = 64) | 7.2 (1.41)
  1 hour after first dose (n = 64) | 3.6 (1.77)
  prior to second dose: number analyzed (Participants) | 63
  prior to second dose | 7.3 (1.59)
  1 hour after second dose: number analyzed (Participants) | 63
  1 hour after second dose | 4.7 (2.09)
  prior to third dose: number analyzed (Participants) | 58
  prior to third dose | 7.2 (1.6)
  1 hour after third dose: number analyzed (Participants) | 57
  1 hour after third dose | 6.1 (2.71)
  prior to fourth dose: number analyzed (Participants) | 54
  prior to fourth dose | 6.6 (2.21)
  1 hour after fourth dose: number analyzed (Participants) | 54
  1 hour after fourth dose | 4.1 (2.96)
  prior to fifth dose: number analyzed (Participants) | 53
  prior to fifth dose | 4.9 (2.57)
  1 hour after fifth dose: number analyzed (Participants) | 53
  1 hour after fifth dose | 2.7 (2.47)
  prior to sixth dose: number analyzed (Participants) | 53
  prior to sixth dose | 4.5 (2.35)

25. Secondary Outcome: Mean Pain Intensity Scores at Relative Time - Matching Placebo Randomized Participants
Description: as for outcome 24
Time Frame: Baseline; for the first 6 administrations
Population: Participants contributing data (indicated in brackets)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Matching Placebo Intravenous: Matching Placebo will be given by intravenous infusion. Matching Placebo will be administered every 4 hours. Ibuprofen 600 mg orally may be given as rescue medication for pain not controlled by Tapentadol alone.
Arm/Group | Matching Placebo Intravenous
Number analyzed (Participants) | 65
units on a scale
  Prior to first dose | 7.3 (1.54)
  1 hour after first dose: number analyzed (Participants) | 64
  1 hour after first dose | 7.8 (1.76)
  prior to second dose: number analyzed (Participants) | 63
  prior to second dose | 8.4 (1.30)
  1 hour after second dose: number analyzed (Participants) | 63
  1 hour after second dose | 8.6 (1.53)
  prior to third dose: number analyzed (Participants) | 23
  prior to third dose | 7.9 (1.65)
  1 hour after third dose: number analyzed (Participants) | 23
  1 hour after third dose | 7.9 (1.77)
  prior to fourth dose: number analyzed (Participants) | 19
  prior to fourth dose | 7.3 (2.05)
  1 hour after fourth dose: number analyzed (Participants) | 19
  1 hour after fourth dose | 7.1 (2.07)
  prior to fifth dose: number analyzed (Participants) | 15
  prior to fifth dose | 5.8 (2.04)
  1 hour after fifth dose: number analyzed (Participants) | 15
  1 hour after fifth dose | 5.2 (2.24)
  prior to sixth dose: number analyzed (Participants) | 15
  prior to sixth dose | 5.7 (2.13)
  1 hour after sixth dose: number analyzed (Participants) | 15
  1 hour after sixth dose | 4.8 (1.76)

ADVERSE EVENTS:
Time Frame: From administration of first dose of study drug up to 4 days after the administration of the last dose of study drug.
Arm/Group | Tapentadol Intravenous | Matching Placebo Intravenous
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/65
Other Adverse Events (participants affected / at risk) | 63/64 | 37/65
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol Intravenous (N=64) | Matching Placebo Intravenous (N=65)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0
Chest discomfort (General disorders) | 1 | 0
Chills (General disorders) | 2 | 0
Cognitive disorder (Nervous system disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 3 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 25 | 8
Dry mouth (Gastrointestinal disorders) | 6 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Feeling abnormal (General disorders) | 3 | 0
Feeling hot (General disorders) | 13 | 1
Feeling jittery (General disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematocrit decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Headache (Nervous system disorders) | 9 | 2
Helicobacter infection (Infections and infestations) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 11 | 2
Hypertension (Vascular disorders) | 0 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Infusion site erythema (General disorders) | 1 | 0
Infusion site extravasation (General disorders) | 5 | 1
Infusion site phlebitis (General disorders) | 9 | 0
Injection site extravasation (General disorders) | 1 | 0
Injection site induration (General disorders) | 1 | 0
Injection site phlebitis (General disorders) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Local swelling (General disorders) | 1 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 2 | 0
Myoclonus (Nervous system disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 43 | 27
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Nightmare (Psychiatric disorders) | 2 | 0
Nystagmus (Nervous system disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oxygen saturation decreased (Investigations) | 11 | 0
Pain (General disorders) | 1 | 0
Pallor (Vascular disorders) | 0 | 2
Palpitations (Cardiac disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Pharyngeal hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 4
Pyrexia (General disorders) | 1 | 1
Pyuria (Renal and urinary disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Red blood cell count decreased (Investigations) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 27 | 2
Tachycardia (Cardiac disorders) | 0 | 2
Tongue injury (Injury, poisoning and procedural complications) | 0 | 1
Tremor (Nervous system disorders) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Vessel puncture site haematoma (General disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 29 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves the right to review any publication pertaining to the trial before it is submitted for publication. Neither party has the right to prohibit publication unless publication can be shown to affect possible patent rights.